CLINICAL TRIAL: NCT01410877
Title: Assessment of Inspiratory Profiles Through Airflow Resistances Designed to Mimic Inhalers
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM13708
Record Dates: First submitted 2011-08-01; First posted 2011-08-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inhaler naive healthy volunteers

SUMMARY:
It is hypothesized that different inhalation profiles (inhalation flow rate versus time curves) result from different forms of patient training. Furthermore, significant inter-subject variability in these profiles should exist that can, under some circumstances, depend on the design of different inhalation devices; this is because dry powder inhalers have different airflow resistances. The investigators also hypothesize that the spread of flow rate versus time profiles for inhalation can be collected. Finally, these profiles can be analyzed from a group of human subjects and used to define a mean and statistical range of inhalation flow rate versus time curves.

The investigators propose to collect the inhalation profiles from 20 'inhaler naïve' healthy volunteers after they have (a) read a typical inhaler package insert and (b) been formally trained in inhaler use by a pharmacist. No drug exposure will occur. The data will be used from this pilot study to (a) show the inter-subject variability in the inhalation profiles used by adults inhaling through realistic airflow resistances (like those in inhalers) following different types of training (b) show how formal training changes inhalation technique and (c) provide a database of typical inspiratory profiles for use and improvement of realistic tests of inhalers in the laboratory. Since pulmonary deposition from inhalers greatly depends upon the way patients inhale through them, this research will result in a database to improve the design and in vitro characterization of inhalers.

ELIGIBILITY:
* Must be healthy as determined by a health questionnaire
* Must not be currently pregnant (self reported)
* Must not have symptoms of an obstructive or restrictive lung disease or be suffering from allergies or congestion at the time of testing
* Must have Forced 'Expiratory Volume in one second' >'Lower Limit of Normal' predicted
* Must be medically stable with no evidence of acute medical or psychiatric illness,
* Must have never used or been trained to use a dry powder inhaler,
* Must not be currently using any inhaler, nasal spray or drug known to affect lung function, Bronchodilators and decongestants in any form are excluded
* Must be at least 4 feet 10 inch tall,
* Must weigh at least 110 pounds (50 kilograms) and be no more than 264 pounds (120 kilograms)
* Must not currently, or in the past year, have used tobacco products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Greater Richmond Area, Virginia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in inhalation flow rate and inhalation volume after the formal training in use of inhaler | 1 year
  Inhalation Profiles will be collected through different airflow resistance, before and after formal training

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Byron, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, School of Pharmacy, Richmond, Virginia, United States